CLINICAL TRIAL: NCT06240299
Title: Neurofeedback for Nociplastic Pain in Rheumatoid Arthritis
Brief Title: Neurofeedback for Nociplastic Pain in Rheumatoid Arthritis (NECTAR)
Acronym: NECTAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UGN23NE390
Record Dates: First submitted 2023-12-06; First posted 2024-02-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis; Chronic Widespread Pain
MeSH Terms: conditions — Arthritis, Rheumatoid; Chronic Pain | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rheumatoid Arthritis - neurofeedback training (Experimental): Intervention: visual neurofeedback
  Research Assessments
  * EEG: relaxed state and motor imagery
  * Quantitative sensory testing
  Questionnaires (after each intervention session):
  * visual analog scale - rate pain intensity
  * pain description and pain intensity reporting
  * mental strategies, affects (emotional experience) and sensations during NF
  * adverse event reporting
  * NASA task load index
  Questionnaires (week before and week after intervention weeks)
  * Routine Assessment of Patient Index Data 3 (RAPID3)
  * American College of Rheumatology Fibromyalgia Scale (ACRFS)
  * McGill Pain Questionnaire
  * Patient-Reported Outcomes Measurement Information System (PROMIS) Depression
  * PROMIS-Anxiety
  * PROMIS-Fatigue
  * PROMIS-Sleep related impairment
  * Pain Number Rating Scale
  * Generalised Self-Efficiency Scale questionnaire
  * Multidimensional Health Locus of Control Scale questionnaires
  Remote follow-up: semi-structured interview over the telephone
  Interventions: Procedure: Neurofeedback

INTERVENTIONS:
Procedure: Neurofeedback — A noninvasive method based on the voluntary modulation of brain activity, with feedback provided through a graphical user interface shown on a computer screen

SUMMARY:
Rheumatoid arthritis is an autoimmune condition, causing inflammation and pain. Yet pain may persist even when inflammation has been treated. This residual pain, called nociplastic pain, has symptoms of a chronic pain condition called fibromyalgia. There are few effective therapies to address this residual pain. Published literature shows that fibromyalgia can be treated by neurofeedback, a noninvasive method that is based on the voluntary modulation of cortical activity. In this pilot study, the investigators want to test the effect of neurofeedback on the fibromyalgia component of pain in rheumatoid arthritis, and also to investigate its effects on related symptoms such as fatigue and sleep disturbance.

DETAILED DESCRIPTION:
Study Schedule For each participant, the intervention paradigm consists of a 1-week diary of pain, sleep and fatigue prior to baseline assessment, 10 intervention sessions 2-3 times per week, post-intervention assessment and remote post-intervention follow-up interview, one month after the last intervention. Hence, each participant will be enrolled in the study for 11-13 weeks, including the follow-up assessment. In case of short-term health problems (e.g., Covid 19, flu, seasonal allergy, etc), experimental sessions can be postponed for up to one week. A maximum of two sessions can be missed otherwise participants will be withdrawn from the study.

Intervention EEG will be recorded with one unit (16 channels) of a modular EEG device (usbamp, Gtec, Austria) requiring 5-10 min setup. Before neurofeedback training (NF), daily baseline EEG activity will be recorded for 2 min, during which participants will sit in a relaxed state, with eyes open. After that, participants will see a graphical user interface (GUI) consisting of three bars that correspond to signal power in three frequency bands: theta, alpha and beta. The bars change colour and height proportionally to the band power. Participants will be aiming to decrease theta and beta and to increase alpha band power as compared to the baseline values. If the power of a particular band passes the threshold level set by the daily baseline recording, the corresponding column turns green, otherwise, the colour is red. NF will be provided from the sensorimotor cortex (electrode locations C4/C3). In total, each training session lasts for 30 min. A second, 2min long EEG recording in the relaxed state with eyes opened will be recorded immediately after the NF session. The experimenter will advise participants on successful mental strategies in the first 3 sessions and will let participants choose their preferred strategy during sessions 4-10.

Baseline EEG recording Participants will be comfortably sitting approximately 1 meter from a computer screen. EEG will be recorded with 4 units (64 channels, passive electrodes) of modular multichannel EEG. This setup requires up to 30 min. EEG will be recorded for 8 min in alternative 2 min blocks of relaxed eyes open and eyes closed state. During eyes open recording, they will be asked to look at a cross in the centre of the screen to avoid excessive eye movements. Following this, participants will be asked to perform cue-based motor imagination practice, i.e., to imagine moving their left and right hands and feet every time they see a cue on a computer screen. Cues will appear in semi-random order, each cue appearing 60 times. A total of 180 trials will be split in six sub-sessions, each totalling 30 trials (10 right hand, 10 left hand, 10 feet).

Quantitative Sensory Testing Quantitative Sensory Testing (QST) is a standardised methodology to study pain sensitivity in humans. A QST protocol includes a series of noxious and non-noxious stimuli delivered to a patient, followed by a semi-objective method for the patient to rate their perception of each stimulus. In this study, participants will complete an abbreviated QST battery to characterise pain sensitivity. All participants who consent to this procedure will undergo familiarisation training prior to data collection to reduce QST-related anxiety. QST comprise of pressure pain sensitivity test and cuff algometry test. Pressure pain sensitivity (15-20 minutes) will be assessed using a digital algometer with a 1 cm2 rubber probe to quantify pressure pain thresholds (PPT) at multiple body sites. Pressure will be manually increased up to 1000 kilo Pascals (kPa). Cuff algometry (10 minutes) will be used to measure deep muscle tonic pain. This consists of a computer controlled air compressor which delivers varying degrees of pressure to a Velcro-adjusted cuff applied to one gastrocnemius muscle.

Visit 1 (week 0): Screening, Consent, Baseline EEG , Questionnaires and Research assessments (including QST). The total duration of Visit 1 will be 4-5 hours including comfort breaks and time for EEG setup.

Visits 2-11 (weeks 1-5): Neurofeedback sessions 1-10, Pain questionnaires (structured and semi-structured). The study visit, including EEG setup (time to put it on and off), intervention and debriefing will take 60-70 min.

Visit 12 (week 6): post-intervention EEG, Questionnaires and Research assessments (including QST). This assessment will take place within 7 (±5) days after the last NF session. The total duration of Visit 12 will be 4-5 hours including comfort breaks and time for EEG setup.

Visit 13 (week 10): remote follow-up. A 10 min semi-structured interview, covering topics such as pain, sleep, fatigue and any adverse effects. The interview will take place over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilment of the ACR/EULAR Classification Criteria for rheumatoid arthritis (RA)
* Fulfilment of the American College of Rheumatology criteria for chronic widespread pain
* Stable disease (swollen joint count ≤1 and CRP ≤10)
* Has normal or corrected to normal vision and hearing abilities
* Right-handed (to reduce baseline motor response test heterogeneity)
* Pain intensity equal or larger than 4 on the Visual Numerical Scale (0 no pain, 10, max pain imaginable)

Exclusion Criteria:

* Unable to understand the task.
* Unable to provide a written informed consent.
* Unable to understand English.
* Major confounding neurological diseases including Multiple Sclerosis, Stroke, Traumatic Brain Injury, Parkinson's Disease, and Alzheimer's Disease)
* Medical or psychiatric conditions that in the judgment of study personnel would preclude participation in the study (psychosis, suicidal ideation etc)
* Under active management of pain team (changing medications, other non pharmacological pain treatment)
* Involved in other interventional experimental studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Difference in nociplastic pain (Visual Analog Scale) | 4 weeks
  Difference in nociplastic pain following 10 sessions of neurofeedback, compared to baseline, as measured by a on a 10 point Visual Analog Scale (VAN), from 1 to 10, where 10 is the highest possible pain. Improvement is indicated by a reduction in score.

SECONDARY OUTCOMES:
Difference in nociplastic pain (ACRFS) | 5 weeks
  Difference in nociplastic pain following 10 sessions of neurofeedback, compared to baseline, as measured by the American College of Rheumatology Fibromyalgia Scale (ACRFS). The score ranges between 0-19, with improvement indicated by a reduction in score.
Difference in nociplastic pain (ACRFS) 1 month post-intervention | 10 weeks
  Difference in nociplastic pain 1 month after the last session, compared to baseline, as measured by the American College of Rheumatology Fibromyalgia Scale (ACRFS). The score ranges between 0-19, with improvement indicated by a reduction in score.
Success of performing neurofeedback | 5 weeks
  EEG power in theta (4-8 Hz), alpha (8-12 Hz) , low beta (13-20 Hz), high beta (20-30) and gamma (30-45 Hz) during NF compared to daily baseline, to assess the success of performing neurofeedback
Mental strategies during neurofeedback | 5 weeks
  Self-reported mental strategies (a goal-directed mental action performed in order to control the graphical user interface) and affects (emotional experience e.g.happy, excited, frustrated, anxious etc.) during NF
Multidimensional Health Locus of Control Scale | 6 weeks
  Questionnaire that evaluates the quality of life in patients with diseases or disabilities, containing 18 questions or statements. For each statement, the participant rates their level of agreement on a 6 point scale, from strongly disagree, to strongly agree.
NASA task load index | 5 weeks
  Questionnaire that rates perceived workload in order to assess the neurofeedback task. The participant rates, on a 20-point visual scale, each of the following aspects: mental demand, physical demand, temporal demand, performance, effort and frustration. Higher scores represent a higher task workload.
7-Day Symptom Diary | 5 weeks
  Pain severity following 10 NF sessions (as measured by 7-Day Symptom Diary (Number Rating Scale between 0-10). A reduction in score represents better outcome.
McGill Pain Questionnaire | 6 weeks
  Multidimensional pain questionnaire. Different types of pain are rated from 0-3 (none to severe pain). A reduction in score represents better outcome.
Self-report of adverse events | 5 weeks
  Adverse events self-report after each NF session

CONTACTS AND LOCATIONS:
Overall Officials: Neil Basu, MD, PhD, Principal Investigator — NHS Greater Galsgow and Clyde
Locations (1):
- Clinical Research Facility (CRF), Queen Elizabeth University Hospital, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Shared on request
Supporting Information: Study Protocol
Time Frame: After study end
Access Criteria: Data will be shared upon reasonable request